CLINICAL TRIAL: NCT05356403
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled 12-Week Study to Evaluate the Safety and Efficacy of Oral Difelikefalin in Advanced Chronic Kidney Disease Subjects With Moderate-to-Severe Pruritus With an up to 52-Week Long-term Extension
Brief Title: CR845-310302: A Study to Evaluate the Safety and Efficacy of Difelikefalin in Advanced Chronic Kidney Disease Patients With Moderate-to-Severe Pruritus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Corporate decision to discontinue work in advanced chronic kidney disease
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR845-310302
Record Dates: First submitted 2022-04-18; First posted 2022-05-02 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Chronic Kidney Diseases; Pruritus
Keywords: difelikefalin; CR845; Pruritus; Chronic Itch; Itch; Itching; uremic pruritus; CKD; CKD-aP; CKD-associated pruritus; Chronic Kidney Disease; Kidney dysfunction; Generalized pruritus; Hemodialysis; Dialysis; ESRD (end stage renal disease); Kidney failure, chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic; Pruritus; Kidney Failure, Chronic | interventions — difelikefalin; Tablets

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled study
Who Masked: Participant, Investigator
Masking Description: Difelikefalin and placebo will be provided as enteric-coated tablets. All tablets are white in color with no markings and are identical in appearance. Difelikefalin tablets will be provided at doses of 1 mg.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Difelikefalin 1 mg Oral Tablet (Experimental): Patients receive oral difelikefalin 1 mg once daily
  Interventions: Drug: Difelikefalin 1 mg Oral Tablet
- Placebo Oral Tablet (Placebo Comparator): Patients receive oral placebo once daily
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Difelikefalin 1 mg Oral Tablet — Difelikefalin 1 mg medication taken orally 1 time/day
  Other Names: CR845
  Arms: Difelikefalin 1 mg Oral Tablet
Drug: Placebo Oral Tablet — Placebo tablet taken orally 1 time/day
  Arms: Placebo Oral Tablet

SUMMARY:
This is a multicenter, double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy of oral difelikefalin administered as a 1 mg tablet once daily compared to placebo in reducing the intensity of itch in advanced chronic kidney disease (CKD) patients with moderate-to-severe pruritus. This study is comprised of an Efficacy Assessment Phase and a Long-term Extension Phase. The Efficacy Assessment Phase includes a double-blind 12-week Treatment Period (Treatment Period 1), and the Long-term Extension Phase includes a double-blind Treatment Period (Treatment Period 2) of up to 52 weeks.

DETAILED DESCRIPTION:
This study will consist of a Screening Period, a 7-day Run-in Period, a 12 week double-blind Efficacy Assessment Phase (Treatment Period 1), a double-blind Long-term Extension Phase (Treatment Period 2) of up to 52 weeks, and a Follow-up Visit (7 to 10 days after the End of Treatment (EOT)/Early Termination (ET) Visit).

If patients continue to meet all inclusion and no exclusion criteria at the end of the 7-day Run-in Period, they will be randomized in a 1:1 ratio to receive once daily oral difelikefalin tablets at a dose of 1 mg or placebo for 12 weeks. Subjects will be stratified according to their use or nonuse of medications to treat pruritus prior to randomization as well as the presence or absence of specific medical conditions. During the Long-term Extension Phase, patients will be re-randomized on Day 1 of Treatment Period 2 to receive either oral difelikefalin 1 mg or placebo, once daily for up to an additional 52 weeks. A final safety Follow-up Visit will be conducted 7 to 10 days after the EOT/ET.

Informed consent will be obtained prior to performing any study-specific procedures. Screening will occur within 7 to 28 days prior to randomization to assess eligibility.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion into the study, a patient must meet the following criteria:

* Advanced stage 4 and 5 CKD and end stage renal disease on hemodialysis
* Subject self-reports experiencing at least near-daily (eg, most days of a week) pruritus for at least 6 months prior to screening.
* Inadequate response to current or prior treatments (including emollients/moisturizers, topical medications, or systemic treatments) for pruritus prior to screening.

Prior to randomization on Day 1 of Treatment Period 1:

1. Has recorded at least 4 WI-NRS scores during the 7-day Run-in Period; and
2. Has a mean baseline WI-NRS score ≥ 5, defined as the average of all non-missing scores reported during the 7-day Run-in Period.

Exclusion Criteria:

A patient will be excluded from the study if any of the following criteria are met:

* Scheduled to receive a renal replacement therapy (dialysis or kidney transplant) during the study.
* Has a concomitant disease, significant medical condition or physical/laboratory/ECG/vital signs abnormality that, in the opinion of the investigator, puts the subject at undue risk or interferes with interpretation of study results, impedes completion of the study procedures, or compromises the validity of the study measurements.
* New or change of treatment received for itch, including antihistamines and corticosteroids (oral, intravenous, or topical), within 14 days prior to the start of run-in.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Efficacy Assessment Phase (Treatment Period 1): Proportion of subjects achieving at least a 4-point improvement from baseline with respect to the weekly mean of the daily 24-hour WI-NRS score at Week 12 of Treatment Period 1 | Week 12 of Treatment Period 1
  Intensity of itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable".

SECONDARY OUTCOMES:
Efficacy Assessment Phase (Treatment Period 1): Proportion of subjects achieving at least a 4-point improvement from baseline with respect to the weekly mean of the WI-NRS at Week 8 of Treatment Period 1. | Week 8 of Treatment Period 1
  Intensity of itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable".
Efficacy Assessment Phase (Treatment Period 1): Proportion of subjects achieving at least a 4-point improvement from baseline with respect to the weekly mean of the WI-NRS at Week 4 of Treatment Period 1. | Week 4 of Treatment Period 1
  Intensity of itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable".
Efficacy Assessment Phase (Treatment Period 1): Proportion of subjects who are "complete itch responders" defined as subjects with ≥ 70% of the non-missing 24-hour WI-NRS scores equal to 0 or 1 at Week 12 of Treatment Period 1. | Week 12 of Treatment Period 1
  Intensity of itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable".
Efficacy Assessment Phase (Treatment Period 1): Change from baseline in Sleep Quality Questionnaire score at the end of Week 12 of Treatment Period 1. | Week 12 of Treatment Period 1
  Sleep Quality will be measured using an NRS used to indicate how much itch has interfered with sleep during the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "did not interfere" and "10" represents "completely interfered".

CONTACTS AND LOCATIONS:
Overall Officials: Cara Therapeutics, PhD, Study Director — Cara Therapeutics
Locations (72):
- United States (8):
  - Cara Therapeutics Study Site, Northridge, California
  - Cara Therapeutics Study Site, Miami, Florida
  - Cara Therapeutics Study Site, Miami Lakes, Florida
  - Cara Therapeutics Study Site, Weston, Florida
  - Cara Therapeutics Study Site, Brunswick, Georgia
  - Cara Therapeutics Study Site, New York, New York
  - Cara Therapeutics Study Site, Orangeburg, South Carolina
  - Cara Therapeutics Study Site, Sugar Land, Texas
- Argentina (6):
  - Cara Therapeutics Study Site, Ciudad Autonoma de Buenos Aire
  - Cara Therapeutics Study Site, Corrientes
  - Cara Therapeutics Study Site, Lanús
  - Cara Therapeutics Study Site, Mar del Plata
  - Cara Therapeutics Study Site, San Nicolás
  - Cara Therapeutics Study Site, Sarandí
- Australia (10):
  - Cara Therapeutics Study Site, Adelaide
  - Cara Therapeutics Study Site, Camperdown
  - Cara Therapeutics Study Site, Concord
  - Cara Therapeutics Study Site, Gosford
  - Cara Therapeutics Study Site, Kogarah
  - Cara Therapeutics Study Site, Launceston
  - Cara Therapeutics Study Site, Liverpool
  - Cara Therapeutics Study Site, Melbourne
  - Cara Therapeutics Study Site, Saint Albans
  - Cara Therapeutics Study Site, Westmead
- Brazil (7):
  - Cara Therapeutics Study Site, Belo Horizonte
  - Cara Therapeutics Study Site, Joinville
  - Cara Therapeutics Study Site, Salvador
  - Cara Therapeutics Study Site, São Bernardo do Campo
  - Cara Therapeutics Study Site, São José do Rio Preto
  - Cara Therapeutics Study Site, São Paulo
  - Cara Therapeutics Study Site 2, São Paulo
- Bulgaria (4):
  - Cara Therapeutics Study Site, Dobrich
  - Cara Therapeutics Study Site, Gabrovo
  - Cara Therapeutics Study Site, Montana
  - Cara Therapeutics Study Site, Plovdiv
- Germany (2):
  - Cara Therapeutics Study Site, Heilbronn
  - Cara Therapeutics Study Site, Kaiserslautern
- Hungary (4):
  - Cara Therapeutics Study Site, Baja
  - Cara Therapeutics Study Site, Budapest
  - Cara Therapeutics Study Site, Kistarcsa
  - Cara Therapeutics Study Site, Pécs
- Italy (4):
  - Cara Therapeutics Study Site, Florence
  - Cara Therapeutics Study Site, Modena
  - Cara Therapeutics Study Site, Pavia
  - Cara Therapeutics Study Site, Roma
- Mexico (4):
  - Cara Therapeutics Study Site, Aguas Calientes
  - Cara Therapeutics Study Site, Durango
  - Cara Therapeutics Study Site, Guadalajara
  - Cara Therapeutics Study Site, Mérida
- Poland (7):
  - Cara Therapeutics Study Site, Golub-Dobrzyń
  - Cara Therapeutics Study Site, Katowice
  - Cara Therapeutics Study Site 2, Krakow
  - Cara Therapeutics Study Site, Krakow
  - Cara Therapeutics Study Site, Lodz
  - Cara Therapeutics Study Site, Szczecin
  - Cara Therapeutics Study Site, Wroclaw
- Romania (3):
  - Cara Therapeutics Study Site, Bucharest
  - Cara Therapeutics Study Site, Oradea
  - Cara Therapeutics Study Site, Timișoara
- South Korea (4):
  - Cara Therapeutics Study Site, Daegu
  - Cara Therapeutics Study Site 2, Goyang-si
  - Cara Therapeutics Study Site, Goyang-si
  - Cara Therapeutics Study Site, Seoul
- Spain (9):
  - Cara Therapeutics Study Site, Almería
  - Cara Therapeutics Study Site, Badalona
  - Cara Therapeutics Study Site, Barcelona
  - Cara Therapeutics Study Site, Ferrol
  - Cara Therapeutics Study Site, Madrid
  - Cara Therapeutics Study Site, Palma de Mallorca
  - Cara Therapeutics Study Site 2, Valencia
  - Cara Therapeutics Study Site, Valencia
  - Cara Therapeutics Study Site, Vitoria-Gasteiz

IPD SHARING:
Plan to Share IPD: No